CLINICAL TRIAL: NCT06112964
Title: Understanding the Impact on CANcer on Neurobehavioral Mechanisms and COGnition in Cachexia (CANCOG)
Brief Title: Neurobehavioural and Cognitive Changes in Cancer Cachexia (CANCOG)
Acronym: CANCOG
Status: Recruiting | Type: Observational
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Dr Anthony Coll, University Associate Professor, University of Cambridge
Other Study IDs: A096708
Record Dates: First submitted 2023-10-24; First posted 2023-11-02 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Cancer; Cachexia; Cachexia-Anorexia Syndrome; Appetite Loss; Weight Loss
MeSH Terms: conditions — Neoplasms; Cachexia; Anorexia; Weight Loss | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — A 10-20ml blood sample will be collected from participants and stored for possible future batch analysis of analytes considered relevant to metabolism, nutrition, body composition, neuro-behaviour or appetite control,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with cancer and cancer associated weight loss/ loss of appetite: Participants with confirmed malignancy, reporting weight loss of >5% body weight in 6 months, or loss of appetite.
  Interventions: Procedure: MRI/ Functional MRI; Behavioral: Self-reported questionnaires; Behavioral: Computer based tasks
- Healthy volunteers: No malignancy or weight loss in the past 6 months
  Interventions: Procedure: MRI/ Functional MRI; Behavioral: Self-reported questionnaires; Behavioral: Computer based tasks

INTERVENTIONS:
Procedure: MRI/ Functional MRI — Participants will undergo an MRI scan lasting approximately 1 hour to examine the structure and function of the brain. During the scan, they will also be asked to perform computer based tasks. This is called functional MRI.
Behavioral: Self-reported questionnaires — Participants will complete questionnaires covering subjective measures relating to food attitudes and intake, and report-based measures of relevant psychopathology including depression and anxiety. These will be derived from standardised scales already used clinically, including the setting of eating disorders and normative studies of the neuroscience of appetite.
Behavioral: Computer based tasks — Participants will complete computer based tasks which are focused specifically on aspects of appetite-related and reward behaviours. Typically, such behaviours are characterised under the following sub-headings:
  i) Motivation (the amount of effort, cognitive or physical, that a person is prepared to expend in order to gain access to food), ii) Valuation (the relative rating of foods in comparison to each other and to non-food items), and iii) Hedonic response (the subjective pleasure experienced in consumption) to food intake

SUMMARY:
The goal of this observational study is to to look for changes within the brain, and changes in body-to-brain signals in people with cancer and people who do not have cancer. The main questions it aims to answer are:

1. Are there differences in areas of the brain known to be related to appetite control, food reward and motivation, between participants with cancer related weight loss and healthy volunteers
2. Do responses to questionnaires and computer based tasks suggest participants with cancer related weight loss have reduced appetite and reduced motivation to eat compared to healthy volunteers, and if so, do questionnaires suggest that this is associated with any other symptoms?

Researchers will compare the structure and blood flow in relevant areas of the brain using MRI images between participants with cancer related weight loss and healthy volunteers. Participants will complete questionnaires and computer based tasks to allow researchers to assess areas of the brain which become more active in response to different stimuli. Some computer based tasks will be performed during the MRI scan. This is called functional MRI.

A further objective is to obtain an archive of blood samples which will be stored securely for future analysis if relevant hormones or analytes are identified that may be relevant to metabolism or body composition

DETAILED DESCRIPTION:
Cancer cachexia is a complex disorder involving progressive loss of muscle and fat in people with cancer, which cannot be corrected with dietary supplements. It affects 50-80% of the cancer population, and accounts for up to 20% of cancer related deaths.To date there are no effective treatments for cancer cachexia and further research is needed to highlight possible treatments for this condition.

Previous research into conditions such as obesity and anorexia have shown the importance of signals between the body and the brain in controlling appetite. This study will focus on how cancer affects signals within the body which are communicated to the brain. In people with cancer, these signals may be altered, leading to changes in appetite and less pleasure from eating, ultimately resulting in weight loss (cancer cachexia).

The study will be observational and will be carried out in one centre at the Translational Research Facility, Addenbrookes Hospital. Researchers aim to recruit 50 participants (30 with cancer and weight loss, and 20 healthy volunteers).

Potential participants will be identified by clinical teams in oncology clinics, via recruitment posters and multi-disciplinary team meetings on the hospital site. Participants will attend for one study visit lasting 4 hours. During this time, participants will undergo an MRI scan, complete questionnaires and perform computer based tasks. Researchers will look for changes within the brain, and changes in body-to-brain signals in people with cancer and people who do not have cancer. Researchers will assess attitudes to eating and body perceptions using questionnaires and computer based tasks. This will indicate whether cancer is driving changes in behaviour which may cause weight loss (cachexia). The ultimate goal is to develop treatment strategies in future to prevent weight loss and improve outcomes for people with cancer

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria for all groups:

* Written informed consent
* Aged 18 years or over
* Willing and able to comply with study procedures and visits

Additional inclusion criteria for participants with cancer:

* Histological or cytological diagnosis of cancer or confirmed non-intracranial malignancy on imaging.
* Unintended documented weight loss of >5% body weight in 6 months which is felt to be cancer related, OR patient reported weight loss and/or change in appetite

Exclusion Criteria:

General exclusion criteria for all groups:

* Non-fluent English speaker
* Active infection, as determined by the investigator based on clinical symptoms and / or fever and / or requirement for antibiotics
* Women, who are pregnant, plan to become pregnant or are lactating.
* MRI contraindication
* A significant acute, chronic or psychiatric condition which in the judgement of the investigator would place the volunteer at undue risk or interfere with the study
* Metabolically or clinically unstable on day of study visit
* Artificial nutrition
* Taking medications which, as determined by the investigator, may affect appetite or cognition, or otherwise affect completion of study tasks.
* Weight or body circumference above upper threshold for MRI scanner (220kg)
* Unresolved obstructive gastrointestinal (GI) lesion

Additional exclusion criteria for participants with cancer:

• Intracranial cancer or metastatic intracranial involvement of cancer

Additional exclusion criteria for healthy volunteers:

* Have, or be recovering from, any form of cancer
* Unintentional weight loss of >5% body weight or unexplained loss of appetite

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A maximum of 50 participants will be recruited to this study over a period of 4 years.
  This will include approximately 30 participants with cancer, and 20 healthy volunteers. Participants with cancer will be recruited from oncology outpatient clinics or multi-disciplinary team meetings including palliative care MDT meetings at Addenbrooke's Hospital, Cambridge. Healthy volunteers will be recruited by advertising on site, study recruitment notice boards or through a contact of the participant with cancer. Participants in each group will be matched for age and sex
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
To characterise structural and functional neuroanatomy as well as neurometabolism through MRI brain imaging in participants with cancer related weight loss and healthy volunteers. | 1 hour
  Eligible participants will undergo an MRI scan during a 1-hour scanning session at Wolfson Brain Imaging Centre.

SECONDARY OUTCOMES:
To determine if there is a difference in food motivation and reward -based behaviour using functional MRI. | 1 hour
  Participants will be asked to perform one computer based task during their MRI scan, which is called functional MRI. Imaging analysis of the results of this task will indicate differences in MRI responses in areas of the brain related to food reward and food motivation, between people with cancer and weight loss and healthy volunteers.
Participants will be asked to perform two computer based tasks after the MRI scan, which have been validated to assess food reward and motivation. | 2 hours
  Participants will be asked to perform two computer based tasks using a laptop. The generated results of these tasks will indicate participants' level of food reward and food motivation and will allow for comparison between people with cancer and weight loss, and healthy volunteers.
To compare responses to questionnaire-based measures of food attitudes, food intake and relevant psychopathology across patients with cancer related weight loss and healthy volunteers. | 1 hour
  The following questionnaires cover food attitudes and intake, and measures of psychopathology including depression and anxiety. These will be derived from standardised scales, used the setting of eating disorders and neuroscience of appetite studies. Questionnaire scores will be compared between people with cancer and weight loss and healthy volunteers.
  Godin Leisure Time Exercise Questionnaire Functional Assessment of Chronic Illness Therapy- Fatigue Functional Assessment of Anorexia/Cachexia Therapy Activities of daily living questionnaire Instrumental activities of daily living scale Scored Patient Generated Subjective Global Assessment Edmonton Symptom Assessment Brief Pain Inventory Patient Health Questionnaire- 9 General Anxiety disorder Hospital Anxiety and Depression Scale Body Perception Questionnaire Snaith Hamilton Pleasure Scale The three factor eating questionnaire DSM-5 Self rated Level 1 Cross-cutting symptom measure
To secure an archive of blood samples for potential future analysis as other targets may become available with research progression locally or within the wider CANCAN consortium | 5 minutes
  A 10-20ml blood sample will be collected from all participants

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Coll, Principal Investigator — University of Cambridge
Locations (1):
- University of Cambridge, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No